CLINICAL TRIAL: NCT05265221
Title: Learning Curve Analysis for Endoscopic Submucosal Dissection of Gastric Neoplasm
Brief Title: Learning Curve for Gastric Endoscopic Submucosal Dissection
Status: Completed | Type: Observational
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Jun-Hyung Cho, Associate Professor, Soonchunhyang University Hospital
Other Study IDs: SCH-ESD-2022
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Endoscopic Submucosal Dissection; Gastric Neoplasm
MeSH Terms: conditions — Stomach Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — All resected specimens were immersed in 10 % formalin. Resected ESD specimens were ﬁxed with pins, then sliced serially at 2-mm intervals, and embedded in a parafﬁn block. If the piecemeal resection was performed, all pieces were reconstructed carefully.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic submucosal dissection — ESD was performed under conscious sedation. For sedation, midazolam and/or propofol were administered intravenously, with cardiorespiratory monitoring. Initially, indigo carmine dye was sprayed onto the tumor to clarify the margin. Then, markings were made 10 mm outside the tumor margin using argon plasma coagulation. After marking, a mixture of sodium hyaluronate with indigo carmine and epinephrine was injected into the submucosa outside the marking dots. Circumferential mucosal incision and submucosal dissection were performed using a Dual and/or IT knife. During the procedure, immediate bleeding was treated by Coagrasper. After ESD, chest and abdominal plain radiography were performed routinely for detection of gastric perforation.

SUMMARY:
Endoscopic submucosal dissection (ESD) for early gastric cancer is a widely accepted treatment option of expanded indication worldwide.

ESD is relatively difﬁcult compared with endoscopic mucosal resection, thus, proper training is essential for the safe performance of the procedure. Thus, it is necessary to receive proper training in the procedure for safe performance of ESD. Previous studies reported that there was a learning curve in ESD training and preceptees needed to perform at least 30-40 procedures in order to master this technique. However, there is few study about the association between the clinical characteristics and competence level for gastric ESD.

DETAILED DESCRIPTION:
This study aims to evaluate the clinical outcomes of ESD and to describe the learning curve for ESD of the gastric neoplasm, based on the analysis of a single endoscopist's experience.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed gastric neoplasm

Exclusion Criteria:

* Age < 20
* History of gastric surgery
* Severe systemic disease
* Advanced chronic liver disease
* Recent history of upper gastrointestinal bleeding

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who underwent endoscopic dissection due to gastric neoplasms
Sampling Method: Non-Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Resection speed | 4 weeks
  Deﬁned as resected lesion size divided by ESD procedure time

SECONDARY OUTCOMES:
Complication rate | 4 weeks
  ESD-related bleeding, gastric perforation, patient's death

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Hyung Cho, M.D., Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- Soonchunhyang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No